CLINICAL TRIAL: NCT03140345
Title: Integrative Nursing Assessment on Hemodialysis Vascular Access
Brief Title: Integrative HD Vascular Access Assessment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Chiang, Hui-Chu, Assistant Professor, National Taipei University of Nursing and Health Sciences
Other Study IDs: TCMG/NTUNHS105-B- 12-02
Record Dates: First submitted 2017-04-16; First posted 2017-05-04 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Renal Dialysis; Integrative Medicine; Hemodialysis Access Failure
Keywords: Hemodialysis; Microcirculation; Traditional Chinese Medicine; Hemodialysis vascular access

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this two-year study is to explore the relationship among function of HVA, nail-fold capillaries and TCM constitutions based on hybridizing data mining techniques. This study will not only improve our understanding on the expressions of function of HVA, nailfold capillaries and tendency of TCM patterns, but also demonstrate the fundamental knowledge of a novel healthcare model on hemodialysis vascular access.

DETAILED DESCRIPTION:
Background

The effectiveness of hemodialysis (HD) depends on HD vascular access (HVA). Individualized prevention based on TCM constitutions can help persons to restore balance and prevent disease. To prevent the negative development of HVA and maintain HVA patency, development of an integrative model of HVA should be an important issue in nephrological nursing. To establish an integrative healthcare model of HVA, the understanding of the relationships between the common TCM constitution patterns of HD patients and the functions of HVA must be improved. In traditional Chinese medicine (TCM), health is conceived as a balance among the elements of the body. Published articles revealed that vascular access surgery, hemodynamic disorder and HD might impact HVA and the microcirculation of HD patients. Hence, changes of hand microcirculation might may come with and indicate the degeneration of HVA.

Purpose

The aims of this two-year study are as follows.

1. To identify major risk factors for the functions of HVA.
2. To measure the microcirculation and constitutions of HD patients.
3. To explore associations among risk factors for the functions of HVA, TCM constitutions and the characteristics of nail-fold capillaries.
4. To propose an HVA assessment model.

Patient

The adult ESRD patients have HD in two hospitals in the north of Taiwan

Data collection

Following approval by the Institutional Review Board, all eligible adult ESRD patients having HD in two hospitals in the north of Taiwan will be invited to participate in the study, after its requirements have been clearly explained to them.

Medical record review, measurements of microcirculation, and TCM constitutions questionnaires, will be used to collect data of eligible patients who provide informed consent.

Demographics, comorbidities, concurrent medication, histories of HVA and HD, parameters related to the adequacy of dialysis, and blood biochemistry data will be retrieved retrospectively from nursing and medical records and entered into a database. The TCM constitution of participants will be measured by questionnaires.

Before dialysis, nail-fold microcirculation will be noninvasively measured using a vediocapillaroscopic device (MC-380, Computed Microcirculation System, Kowa Optics Corp., Taiwan). The equipment and measuring procedures will be explained to the subjects. A finger to be examined will be gently placed on a microscope base plate and held still for the duration of the measurement. Computerized image processing will be used to capture and analyze data. The following morphological data will be extracted: blood velocity, capillary density, capillary width, capillary length, and the presence of abnormal capillary morphology.To identify the common microcirculation patterns of HD patients, images of nail-fold capillary will be processed use a framework that was developed by Prof. K. P. Lin and colleagues.

Statistical analysis

All of the collected data will be entered into a database. The Statistical Package for the Social Sciences for Windows (SPSS Inc, Chicago, Ill) was used to perform statistical analyses. Baseline demographics, comorbidities, medication, the results of blood biochemistry tests, and parameters that are related to HD adequacy and access function are presented as means, standard deviation and proportions as appropriate. Associations between parameters regarding vascular access dysfunction and the other variables were analyzed using the t-test, one-way analysis of variance, and Pearson's correlation coefficients, as appropriate. P<0.05 was considered to indicate statistical significance.

Information regarding the function of HVA will be incomplete if some patients do not experience any HVA dysfunction for the duration of this study. Hence,techniques for censored and truncated data will be used to deal with the incomplete data. Regressions and appropriate survival analysis will be conducted to capture the distribution of the function of HVA, and to identify the independent predictors of HVA function. In this study, a novel hybridizing data mining techniques will be applied to reduce data uncertainty. The HD-index that was developed by Prof. K. Y. Huang will be used to filter out uncertain data and to improve the precision of the forecasting model.

ELIGIBILITY:
Inclusion Criteria:

* having ESRD and needing hemodialysis three times weekly, having undergone hemodialysis ≥ 3 months, speaking Chinese or Taiwanese, and agreeing for data to be collected and stored in a database for analysis

Exclusion Criteria:

* life expectancy ≤ 3 months, having a malignant tumor, having unstable hemodynamics, having had a cerebrovascular accident, having acute heart failure, having acute bronchitis with acute exacerbation, or having had a severe infection in the last three months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult ESRD patients having HD in two hospitals in the north of Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-06-07 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Patency of hemodialysis vascular access | through study completion, an average of 2 year
  Patency of hemodialysis vascular access is defined as 1) the interval from the time of access placement to the time of access abandonment, any patency reestablish intervention, or create new access; and 2) the number of hemodialysis vascular access dysfunction events. The time of access placement and the time of the intervention, as well as number of hemodialysis vascular access dysfunction events will be retrieved from medical records. The interval from the time of access placement to the intervention will be calculated in days.

SECONDARY OUTCOMES:
Nail-fold blood flow velocity of the hands of the paticipants | 2 years
  Nail-fold blood velocity will be measured noninvasively by a vediocapillaroscopic device. The unit of nail-fold blood velocity is um/sec. The difference between two hands and the difference among every measurement will be analyzed.
Total vessel density of nail-fold capillary in the hands of participants. | 2 years
  Total vessel density of nail-fold capillary is the number of capillaries per mm*mm flied. The unit of nail-fold blood velocity is um/sec. The difference between two hands and the difference among every measurement will be analyzed.
Diameter of nail-fold capillary in the hands of participants. | 2 years
  The width of nail-fold capillary in the hand with hemodialysis vascular access will be presented in um. The unit of nail-fold blood velocity is um/sec. The difference between two hands and the difference among every measurement will be analyzed.
Abnormalities of nail-fold capillary in the hands of participants. | 2 years
  The number of microaneurysms, giant capillaries, neoangiogenic capillaries, capillary tortuosity, avascular areas, and hemorrhage will be counted and presented in number/ mm*mm. The unit of nail-fold blood velocity is um/sec. The difference between two hands and the difference among every measurement will be analyzed.
Distribution of the traditional Chinese medicine constitution patterns of HD patients | 8 months
  Proportion of each TCM constitution patterns will be presented while the participants have been measured by the TCM Constitutions Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Chu Chiang, Principal Investigator — College of Nursing
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Jaishi AA, Oliver MJ, Thomas SM, Lok CE, Zhang JC, Garg AX, Kosa SD, Quinn RR, Moist LM. Patency rates of the arteriovenous fistula for hemodialysis: a systematic review and meta-analysis. Am J Kidney Dis. 2014 Mar;63(3):464-78. doi: 10.1053/j.ajkd.2013.08.023. Epub 2013 Oct 30. PMID 24183112
- [Background] Ocak G, Rotmans JI, Vossen CY, Rosendaal FR, Krediet RT, Boeschoten EW, Dekker FW, Verduijn M. Type of arteriovenous vascular access and association with patency and mortality. BMC Nephrol. 2013 Apr 4;14:79. doi: 10.1186/1471-2369-14-79. PMID 23557085
- [Background] Wu CC, Zhang G, Huang TC, Lin KP. Red blood cell velocity measurements of complete capillary in finger nail-fold using optical flow estimation. Microvasc Res. 2009 Dec;78(3):319-24. doi: 10.1016/j.mvr.2009.07.002. Epub 2009 Jul 30. PMID 19647002
- [Background] Wu CC, Lin WC, Zhang G, Chang CW, Liu RS, Lin KP, Huang TC. Accuracy evaluation of RBC velocity measurement in nail-fold capillaries. Microvasc Res. 2011 May;81(3):252-60. doi: 10.1016/j.mvr.2011.01.003. Epub 2011 Jan 19. PMID 21255589